CLINICAL TRIAL: NCT07264374
Title: Comparative Study of Femoral Vein, Internal Jugular Vein and Inferior Vein Cava Collapsibility Indices in Polytrauma Patients Presenting to the Emergency Department by Sonographic Evaluation Before and After Resuscitation.
Brief Title: Femoral Vein, Internal Jugular Vein and Inferior Vein Cava Collapsibility Indices in Polytrauma Patients by Sonographic Evaluation Before and After Resuscitation.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Abdelrady Mahmoud, Comparative Study of Femoral vein, Internal jugular vein and Inferior vein cava Collapsibility Indices in polytrauma patients presenting to the emergency department by sonographic evaluation before and after resuscitation, Assiut University
Other Study IDs: FV-IJV-IVC-CI-shocked-2025
Record Dates: First submitted 2025-10-01; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Shock; Hyopvolemia
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound assesment of FV,IJV and IVC collabsibillity indecis — Ultrasound-Guided Inferior Vena Cava,femoral vein and internal jugular vein collabsibilty indecis Assessment This intervention involves bedside ultrasound measurement of the inferior vena cava (IVC) diameter and calculation of the IVC collapsibility/distensibility index. Assessments will be performed both at initial presentation and after fluid resuscitation in shock patients. The procedure is non-invasive, rapid, and performed according to standardized emergency ultrasound protocols.

SUMMARY:
The aim of this study is to evaluate correlation between the collapsibility indices of the FV or IJV to IVC-CI among polytrauma patients presenting to the ED by sonographic evaluation before and after resuscitation.

DETAILED DESCRIPTION:
Polytrauma patients often present with hemodynamic instability where rapid and accurate assessment of intravascular volume is crucial. Central venous pressure monitoring, though considered a standard, is invasive and not always feasible in emergency settings. Point-of-care ultrasound (POCUS) provides a non-invasive alternative through assessment of venous collapsibility indices.

The inferior vena cava (IVC) collapsibility index is commonly used, but its evaluation may be limited in cases of abdominal trauma, obesity, or technical difficulties. The internal jugular vein (IJV) and femoral vein (FV) are superficial, easily accessible, and may provide reliable alternatives.

This study aims to compare the collapsibility indices of the IVC, IJV, and FV in polytrauma patients before and after resuscitation using sonographic evaluation. The objective is to determine their relative accuracy and feasibility as non-invasive markers of intravascular volume status to guide resuscitation in emergency settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18years. ( Patients presented by hypovolemic shock

Exclusion Criteria:

* Patient refusal Body Mass Index > 40 kg/m2. Cardiac patients or cardiac tamponade Aortic injury or for cardio-thoracic emergent operation Patients with abdominal mass or other pathology as abdominal collection. Any patient needs emergent surgical intervention History of pulmonary artery hypertension. Femoral vein occlusion. Pregnancy. Pulmonary oedema. Patients will need mechanical ventilation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged 18-65 years presenting with shock to the emergency department and requiring volume status assessment through both IVC,FV and IJV collabsibility indecis by ultrasound.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
correlation between the collapsibility indices of the FV or IJV to IVC-CI among polytrauma patients presenting to the ED before and after resuscitation. | correlation between the collapsibility indices of the FV or IJV to IVC-CI among polytrauma patients at time of presentation to the ED and after one hour of resuscitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Emeregency medicine department ,Assiut University, Asyut, Weledea, Egypt